CLINICAL TRIAL: NCT05720260
Title: A Randomized, Phase II Study for Premenopausal Metastatic or Locally Advanced Breast Cancer Patients: Capivasertib, Goserelin, Fulvestrant With/Without Durvalumab, Versus Goserelin, Fulvestrant, and Durvalumab, Versus Goserelin/ Fulvestrant.
Brief Title: Immunotherapy, Hormone Therapy, and AKT Inhibitor for Premenopausal ER Positive MBC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202109031MIPD
Record Dates: First submitted 2023-01-26; First posted 2023-02-09 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-04

CONDITIONS: Premenopausal Breast Cancer; Metastatic Breast Cancer; ER Positive Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Goserelin; Gonadotropin-Releasing Hormone; Fulvestrant; capivasertib; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm A: goserelin/ fulvestrant/ durvalumab (Experimental): Historical control arm (goserelin, fulvestrant) plus immunotherapy
  Interventions: Drug: Goserelin; Drug: Fulvestrant; Drug: Durvalumab
- Arm B: goserelin/ fulvestrant/ capivasertib/ durvalumab (Experimental): Historical control arm (goserelin, fulvestrant) plus AKT inhibitor and immunotherapy
  Interventions: Drug: Goserelin; Drug: Fulvestrant; Drug: Capivasertib; Drug: Durvalumab
- Arm C: goserelin/ fulvestrant/ capivasertib (Experimental): Historical control arm (goserelin, fulvestrant) plus AKT inhibitor and immunotherapy
  Interventions: Drug: Goserelin; Drug: Fulvestrant; Drug: Capivasertib

INTERVENTIONS:
Drug: Goserelin — Hormone therapy
  Other Names: GnRH agonist
Drug: Fulvestrant — Hormone therapy
  Other Names: SERD
Drug: Capivasertib — AKT inhibitor
  Other Names: AZD5363
  Arms: Arm B: goserelin/ fulvestrant/ capivasertib/ durvalumab; Arm C: goserelin/ fulvestrant/ capivasertib
Drug: Durvalumab — immunotherapy
  Other Names: Imfinzi
  Arms: Arm A: goserelin/ fulvestrant/ durvalumab; Arm B: goserelin/ fulvestrant/ capivasertib/ durvalumab

SUMMARY:
This is an open-label randomized phase II study in estrogen receptor positive locally advanced or metastatic breast cancer patients. The main inclusion population are either luminal subtype B by PAM50 analysis or failed less than 2 lines of hormonal therapy for locally advanced or metastatic breast cancer. The subjects have to be premenopausal or perimenopausal and are not allowed to receive any systemic chemotherapy for their locally advanced or metastatic breast cancer. Eligible subjects will be randomized into goserelin/ fulvestrant/ durvalumab (Arm A), goserelin/ fulvestrant/ capivasertib/ durvalumab (Arm B), or goserelin/ fulvestrant/ capivasertib (Arm C) at a 1:1:1 ratio. The primary endpoint is objective response rate (ORR) of the whole other three arm compared to historical goserelin/ fulvestrantcontrol arm. The major secondary endpoint will be progression-free survival or ORR compared among different treatment arms.

DETAILED DESCRIPTION:
This is an open-label randomized phase II study in estrogen receptor positive locally advanced or metastatic breast cancer patients. The main inclusion population are either luminal subtype B by PAM50 analysis or failed less than 2 lines of hormonal therapy for locally advanced or metastatic breast cancer. The subjects have to be premenopausal or perimenopausal and are not allowed to receive any systemic chemotherapy for their locally advanced or metastatic breast cancer. Eligible subjects will be randomized into goserelin/ fulvestrant/ durvalumab (Arm A), goserelin/ fulvestrant/ capivasertib/ durvalumab (Arm B), or goserelin/ fulvestrant/ capivasertib (Arm C) at a 1:1:1 ratio. The primary endpoint is objective response rate (ORR) of the whole other three arm compared to historical goserelin/ fulvestrant control arm. The major secondary endpoint will be progression-free survival or ORR compared among different treatment arms. Secondary endpoints include PFS and ORR comparison between arms. Exploratory endpoints include biomarkers, such as TILs, PD-L1 correlation with treatment response.

ELIGIBILITY:
Inclusion criteria

1. A histological confirmed ER positive (>1%) invasive breast cancer.
2. Locally advanced or metastatic disease with at least one measurable target lesion
3. Patients who had not received chemotherapy for locally advanced or metastatic disease
4. Patients have to be (i) either primary resistant to hormonal therapy defined as recurrence developed within 2 years of adjuvant hormonal therapy (ii) or resistant to prior hormonal therapy (failed ≤ 2lines of hormonal therapy for locally advanced or metastatic breast cancer)
5. Patients must be premenopausal or perimenopausal women according the clinical menstrual history or E2 / FSH level based on local hospital guidance. Patient with menopausal status cannot be determined due to ongoing LHRH agonist treatment is allowed if evidence of premenopausal status prior to patients' LHRH agonist usage can be provided.
6. ECOG 0-1
7. Patients must have adequate organ and marrow reserve measured within 14 days(within screening period ) prior to randomization as defined below:

   * Hemoglobin ≥ 9.0 g/dL;
   * Absolute neutrophil count ≥ 1,500 /L;
   * Platelets ≥ 100,000/L;
   * Total bilirubin ≤ 1.5 x upper normal limit;
   * AST(SGOT)/ALT(SGPT) ≤ 2.5 x upper normal limit; for patients with liver metastases AST(SGOT)/ALT(SGPT) ≤ 5 x upper normal limit is allowed;
   * Serum creatinine ≤ 1.5mg/dL or creatinine clearance ≧50ml/min;
   * aPTT < 1.5 x upper normal limit (unless on therapeutic anti-coagulation);
   * Proteinuria ≤ 1+ with urine dipstick, if > 1+, 24-hour urine protein must be ≤ 1 g.
8. Age older than 20-year-old.
9. All women of childbearing potential must have a negative pregnancy test obtained within 7 days before starting therapy. Patients must not be breastfeeding.
10. Patients with reproductive potential must use effective contraception (hormone or barrier method of birth control) prior to study entry, for the duration of study participation, and for 6 months after the completion of therapy.
11. Patients (or a surrogate) must be able to comply with study procedures and to give signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in the clinical study protocol (CSP). The patients (or a surrogate) must be able to provide of signed and dated written ICF prior to any mandatory study specific procedures, sampling, and analyses.
12. Body weight >30 kg
13. Must have a life expectancy of at least 12 weeks Exclusion criteria

Patients fulfilled ANY of the following criteria will be excluded from this trial:

1. Prior therapy with capivasertib, fulvestrant, anti-PD1 or anti-PDL1 immunotherapy
2. Prior chemotherapy for locally advanced or metastatic breast cancer.
3. Radiotherapy with a wide field of radiation within 4 weeks before the first dose of study treatment
4. The tumor is HER-2 positive by IHC 3+ or IHC 2+/ISH positive.
5. Patients have active brain metastases or spinal cord compression or brain metastases unless asymptomatic, treated and stable and not requiring steroids for at least 4 weeks prior to start of study treatment
6. Other malignancy within 5 years except cured basal cell or squamous cell skin cancer or carcinoma in situ of the cervix.
7. Psychiatric illness or social situation that would preclude study compliance.
8. Serious non-healing wound, ulcer, or bone fracture.
9. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to enrollment.
10. Prior minor surgery within 7 days.
11. History of allergic reaction to compounds of similar chemical composition to the study drugs.
12. Pregnancy or lactation.
13. With the exception of alopecia, any unresolved toxicities from prior therapy greater than CTCAE grade 1 at the time of starting study treatment
14. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C. Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
15. Known to have tested positive for human immunodeficiency virus
16. History of allogenic organ transplantation.
17. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion: a) Patients with vitiligo or alopecia; b) Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement; c)Any chronic skin condition that does not require systemic therapy; d) Patients without active disease in the last 5 years may be included but only after consultation with the study physician; e)Patients with celiac disease controlled by diet alone.
18. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent. Refractory nausea and vomiting, malabsorption syndrome, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection, or other condition that would preclude adequate absorption of capivasertib.
19. History of another primary malignancy except for: a) Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of IP and of low potential risk for recurrence; b) Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease; c)Adequately treated carcinoma in situ without evidence of disease
20. History of leptomeningeal carcinomatosis.
21. Previous allogeneic bone marrow transplant or solid organ transplant.
22. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab. The following are exceptions to this criterion:

    1. Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
    2. Systemic corticosteroids at physiologic doses not to exceed <<10 mg/day>> of prednisone or its equivalent
    3. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
23. Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. Note: Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 30 days after the last dose of IP.
24. Any of the following cardiac criteria at screening:

    * Mean resting corrected QT interval (QTc) >470 msec obtained from 3 consecutive ECGs
    * Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG (eg, complete left bundle branch block, third degree heart block)
    * Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalaemia, potential for Torsades de Pointes, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age or any concomitant medication known to prolong the QT interval
    * Experience of any of the following procedures or conditions in the preceding 6 months: coronary artery bypass graft, angioplasty, vascular stent, myocardial infarction, angina pectoris, congestive heart failure New York Heart Association (NYHA) grade ≥2
    * Uncontrolled hypotension - SBP <90 mmHg and/or DBP <50 mmHg
    * Cardiac ejection fraction outside institutional range of normal or <50% (whichever is higher) as measured by echocardiogram.
25. Clinically significant abnormalities of glucose metabolism as defined by any of the following at screening:

    * Patients with diabetes mellitus type I or diabetes mellitus type II requiring insulin treatment
    * HbA1c ≥8.0% (63.9 mmol/mol)
26. Any investigational agents or study drugs from a previous clinical study within 30 days of the first dose of study treatment
27. Potent inhibitors or inducers of CYP3A4 within 2 weeks prior to the first dose of study treatment (3 weeks for St John's wort), or sensitive substrates of CYP3A4, CYP2C9 and/or CYP2D6 with a narrow therapeutic window within 1 week prior to the first dose of study treatment.
28. Participation in another clinical study with an investigational medicinal product (IMP) administered in the last 30 days or 5 half-lives, whichever is longer
29. History of hypersensitivity to active or inactive excipients of capivasertib, fulvestrant, durvalumab, goserelin or drugs with a similar chemical structure or class to the above-mentioned drugs
30. Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2023-01-17 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | From time of randomization to death or tumor progression whichever comes first in 200 months
  PFS comparison between historical control (fulvestrant and goserelin) and Arm A/B/C

CONTACTS AND LOCATIONS:
Overall Officials: Yen-Shen Lu, MD, PhD, Study Chair — NTUH
Locations (1):
- Department of Oncology, National Taiwan University Hospital, Taipei, Taiwan